CLINICAL TRIAL: NCT01331330
Title: A Clinical Evaluation of Different Device Parameters for the Management of Patients With Treatment Resistant Major Depressive Disorder, Single or Recurrent Episode, With Deep Brain Stimulation
Brief Title: European Deep Brain Stimulation (DBS) Depression Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM-09-035-EU-DB
Record Dates: First submitted 2011-04-04; First posted 2011-04-08 (Estimated); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder; Unipolar; Implantable Stimulation Electrodes
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group B (Active Comparator): Low Programming
  Interventions: Device: Deep Brain Stimulation
- Group A (Experimental): Normal Programming
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Normal DBS Programming
  Arms: Group A
Device: Deep Brain Stimulation — Low Programming
  Arms: Group B

SUMMARY:
To evaluate the effects of two different programming settings of deep brain stimulation (DBS) in the subgenual white matter (Brodmann Area 25 WM) as an adjunctive treatment for treatment resistant Major Depressive Disorder (TR-MDD), single or recurrent episode on mood as measured by the MADRS.

DETAILED DESCRIPTION:
The European Study was a prospective, multicenter, double-blind, randomized study comparing high frequency stimulation (130 Hz) to low frequency stimulation (20 Hz). Subjects underwent 2 baseline evaluations by 2 separate psychiatrists and were implanted with the Libra DBS system. Subjects were randomized to receive either high or low frequency stimulation. The primary endpoint was evaluated after 6 months of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (non-pregnant) age is 21-70 years;
* Diagnosed with non-psychotic major depressive disorder, single or recurrent episode by Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition, Text Revision, 2000 (DSM-IV-TR) criteria derived from the Mini International Neuropsychiatric Interview (MINI);
* First episode onset before age 45;
* Current episode > 12 month duration;
* In the current episode: Documented resistance to a minimum of 4 adequate depression treatments from at least 3 different categories;
* In adult lifetime (>21 year of age) have experience a period of wellness as defined by DSM IV criteria;
* MADRS score ≥22 at 2 separate baseline visits, rated by 2 separate psychiatrists;
* Global Assessment of Functioning (GAF) score <50;
* Mini-mental state examination (MMSE) score >24;
* No change in current antidepressant medication regimen or medication free for at least 4 weeks prior to study entry;
* Able to give informed consent in accordance with institutional policies;

Exclusion Criteria:

* A diagnosis of bipolar I or bipolar II disorder by DSM-IV-TR criteria, derived from the MINI;
* Meets criteria for borderline or antisocial personality disorder in the last 12 months by DSM-IV-TR criteria, derived from the Cluster B Personality Disorders Sections 301.7 - 301.83, preferably screened via Structured Clinical Interview for DSM-IV Personality Disorders (SCID-II) at Baseline visit (optional);
* In the current depressive episode, has been diagnosed with General Anxiety Disorder (GAD) - as defined by the DSM-IV-TR, and GAD is the primary diagnosis;

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott Medical Devices
Locations (5):
- France (2):
  - CHU Pasteur, Nice
  - Hôpital La Pitié Salpêtrière, Paris
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel
- United Kingdom (2):
  - King's College London, London
  - National Hospital for Neurology and Neurosurgery - UCL, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 : High Frequency Group: Group 1 : DBS High Frequency (HF) Group Device Programming (130 Hz) Implanted with investigational device and activated for stimulation.
- Group 2 : Low Frequency Group: Group 2 : DBS Low Frequency (LF) Group Device Programming (20 Hz) Implanted with investigational device and activated for stimulation.
Period: Overall Study
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Started | 5 | 4
Completed | 3 | 3
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Full Range); unit: years] | 43 [33 to 67] | 51 [40 to 64] | 46 [33 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 2 | 4
  Israel | 2 | 2 | 4
  France | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in MADRS Score
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item scale that measures depressive symptom severity. Scores range from 9 to 60, with a higher score indicating more severe depression.
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
percentage change from baseline
  4 months | -7.7 (22.8) | -7.4 (21.9)
  7 months | -8.8 (20.6) | -6.2 (10.1)
  10 months | -42.9 (28.4) | -22.7 (11.4)
  13 months | -37.9 (25.4) | -15.9 (39.1)

2. Secondary Outcome: Mean Percent Change From Baseline in Hamilton Rating Scale for Depression (HDRS) Score
Description: The Hamilton Depression Rating Scale is a 17-item scale that measures depressive symptom severity. Scores range from 0 to 52, with a higher score indicating more severe depression.
Time Frame: 4, 7, 10 and 13 month
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
percent change from baseline
  4 months: number analyzed (Participants) | 5 | 3
  4 months | -6.1 (43.7) | -28.1 (24.3)
  7 months | -3.0 (38.7) | -12.9 (15.6)
  10 months: number analyzed (Participants) | 4 | 2
  10 months | -46.8 (38.4) | -16.5 (3.1)
  13 months: number analyzed (Participants) | 4 | 2
  13 months | -34.5 (35.5) | -21.5 (10.3)

3. Secondary Outcome: Responder Rate (40% Reduction in MADRS)
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
Participants
  4 months: number analyzed (Participants) | 5 | 3
  4 months | 0 | 0
  7 months | 0 | 0
  10 months: number analyzed (Participants) | 4 | 2
  10 months | 3 | 0
  13 months: number analyzed (Participants) | 4 | 2
  13 months | 2 | 1

4. Secondary Outcome: Mean Percent Change From Baseline in Hamilton Anxiety Rating Scale (HAMA-A) Score
Description: Developed by M. Hamilton, this widely-used interview scale measures the severity of a patient's anxiety, based on 14 parameters, including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Group 2 : Low Frequency Group: Group 2 : DBS Low Frequency (LF) Group Device Programming (, 20 Hz)) Implanted with investigational device and activated for stimulation.
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
percentage change from baseline
  4 months | -8.3 (41.0) | -9.5 (50.7)
  7 months | -5.6 (48.0) | -5.9 (31.6)
  10 months | -26.2 (48.9) | -21.9 (6.3)
  13 months | -18.8 (46.1) | 25.1 (62.8)

5. Secondary Outcome: Mean Percent Change From Baseline in GAF Score
Description: The Global Assessment Scale (GAF) is a hypothetical continuum of mental health illness that looks at psychological, social, and occupational functioning. It measures how much a person's symptoms affect their day-to-day life on a scale of 0 to 100. A score of 100-91 indicates no symptoms, 90-81 indicates absent minimal symptoms, 80-71 indicates symptoms that are transient and reactions expectable to psychosocial stressors, 70-61 indicates mild symptoms, 60-51 indicates moderate symptoms, 50-41 indicates serious symptoms, 40-31 indicates some impairment in reality testing or communication OR major impairment in several areas, 30-21 indicates delusions or hallucinations, 20-11 indicates danger of hurting self or others OR occasionally fails to maintain personal hygiene, 10-1 indicates persistent danger of severely hurting self or others OR persistent inability to maintain minimal personal hygiene OR serious suicidal act with clear expectation of death and 0 indicates inadequate data.
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
percentage change from baseline
  4 months | 17.2 (26.4) | 11.1 (19.2)
  7 months | 20.7 (14.8) | 18.5 (17.0)
  10 months | 34.4 (30.7) | 18.8 (26.5)
  13 months | 45.2 (20.9) | 24.3 (18.7)

6. Secondary Outcome: Mean Percent Change From Baseline in Quick Inventory of Depressive Symptoms - Self Report (QIDS-SR) Score
Description: The Quick Inventory of Depressive Symptomatology Self Report (QIDS- SR) is a 16-question shortened self-test, derived from the 30-item Inventory of Depressive Symptomatology (IDS). Questions in the QIDS - SR-116 correlate with the nine Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) symptom criterion domains, Including: Sleep disturbance (initial, middle, and late insomnia or hypersomnia) (Q 1 - 4), Sad mood (Q 5), Decrease/increase in appetite/weight (Q 6 - 9), Concentration (Q 10), Self-criticism (Q 11), Suicidal ideation (Q 12), Interest (Q 13), Energy/fatigue (Q 14), Psychomotor agitation/retardation (Q 15 - 16). The severity of depression can be judged based on the total score. A score of 1-5 indicates No depression, 6-10 indicates Mild depression, 11-15 indicates Moderate depression, 16-20 indicates Severe depression and 21-27 indicates Very severe depression.
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
percentage change from baseline
  4 months | -0.6 (17.1) | -2.8 (38.2)
  7 months | -10.4 (24.6) | -2.3 (13.4)
  10 months | -41.1 (47.2) | -21.0 (36.4)
  13 months | -21.3 (26.7) | -18.7 (33.2)

7. Secondary Outcome: Mean Percent Change From Baseline in Clinical Global Impression of Severity and Improvement (CGI) Severity of Illness
Description: The CGI severity of illness scale is a simple validated, single-item, 7-point self-reported categorical scale ranging from 0-7 where 0 indicates not assessed; 1 indicates normal, not at all ill; 2 indicates borderline mentally ill; 3 indicates mildly ill; 4 indicates moderately ill; 5 indicates markedly ill; 6 indicates severely ill; and 7 indicates among the most severely ill patients.
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
percentage change from baseline
  4 months | -3.5 (20.5) | -6.7 (14.7)
  7 months | -12.6 (13.5) | -12.7 (19.2)
  10 months | -33.6 (16.6) | -8.7 (28.1)
  13 months | -38.6 (15.5) | -8.7 (28.1)

8. Secondary Outcome: Mean Total CGI for Global Improvement Score
Description: The CGI global improvement score ranges from 0-7 where 0 indicates not assessed; 1 indicates very much improved; 2 indicates much improved; 3 indicates minimally improved; 4 indicates no change; 5 indicates minimally worse; 6 indicates much worse; and 7 indicates very much worse.
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
scores on a scale
  4 months | 4.0 (1.6) | 4.0 (1.0)
  7 months | 3.6 (0.5) | 3.3 (0.6)
  10 months | 2.3 (1.3) | 3.0 (0.0)
  13 months | 2.0 (0.8) | 3.5 (0.7)

9. Secondary Outcome: Mean Percent Change From Baseline in Patient Global Impression Index (PGI) Severity of Illness
Description: as for outcome 7
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
percentage change from baseline
  4 months | 11.7 (50.7) | -4.8 (21.6)
  7 months | 12.0 (49.6) | 20.0 (20.0)
  10 months | -26.1 (23.7) | 26.2 (57.2)
  13 months | -24.0 (17) | 26.2 (57.2)

10. Secondary Outcome: Mean Total PGI for Global Improvement Score
Description: as for outcome 8
Time Frame: 4, 7, 10 and 13 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
Number analyzed (Participants) | 5 | 4
scores on a scale
  4 months | 4.2 (1.8) | 4.3 (1.2)
  7 months | 4.0 (1.4) | 4.0 (0.0)
  10 months | 2.3 (1.9) | 4.0 (1.4)
  13 months | 2.3 (1.0) | 3.0 (0.0)

ADVERSE EVENTS:
Arm/Group | Group 1 : High Frequency Group | Group 2 : Low Frequency Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 : High Frequency Group (N=5) | Group 2 : Low Frequency Group (N=4)
Overdose of Diathipin and Valium (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 : High Frequency Group (N=5) | Group 2 : Low Frequency Group (N=4)
Abdominal upset and tremors (Gastrointestinal disorders) | 0 | 1
Abdominal upset, hyperacidity and diarrhea (Gastrointestinal disorders) | 0 | 1
Diarrhea and vomiting (Gastrointestinal disorders) | 0 | 1
Dental abscess (lower jaw on the left side) (General disorders) | 1 | 0
Dizziness and losing balance (otitis media) (General disorders) | 0 | 1
Episode of anxiety (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
First of 2 falls (General disorders) | 0 | 1
Frontal headache on the left side (General disorders) | 0 | 1
Itching at the front hairline (General disorders) | 0 | 1
Itching of the scalp, when the head bandage was on (General disorders) | 0 | 1
Itchy scalp (General disorders) | 0 | 1
Losing balance (General disorders) | 0 | 1
Poor memory to recent events (General disorders) | 0 | 1
Scalp itching under the head bandage (General disorders) | 1 | 0
Second of 2 falls (General disorders) | 0 | 1
Sensation (tingling) in different parts of the face on touching the scalp (General disorders) | 1 | 0
Sore throat, fever, lethargy, drowsiness (General disorders) | 1 | 0
Tightness in the neck (General disorders) | 0 | 1
Blood oozing (bleeding) from the incision on the left side of the scalp (Injury, poisoning and procedural complications) | 0 | 1
Burning sensation over the chest scar (Injury, poisoning and procedural complications) | 1 | 0
Itching and pain at the site of the surgical incision in the chest on moving the left arm (Injury, poisoning and procedural complications) | 1 | 0
Mild headache at the site of the incisions in the scalp (Injury, poisoning and procedural complications) | 0 | 1
Mild pain and tenderness at left upper side of the chest (battery site) (Injury, poisoning and procedural complications) | 0 | 1
Pain (neuralgia) over the left tempromadipular joint and extended to left scalp (Injury, poisoning and procedural complications) | 1 | 0
Pain and tenderness at the site of the chest incision (Injury, poisoning and procedural complications) | 0 | 1
Post operative headache (Injury, poisoning and procedural complications) | 0 | 1
Post surgical headache (mainly in the forehead, throbbing in nature) (Injury, poisoning and procedural complications) | 0 | 1
Redness and mild swelling at the site of the left scalp incision and chest incision (Injury, poisoning and procedural complications) | 0 | 1
Redness and swelling at the site of the chest incision (Injury, poisoning and procedural complications) | 0 | 1
Stabbing pain at the site of the chest surgical incision (Injury, poisoning and procedural complications) | 0 | 1
Tenderness at the left side of the scalp when the patient lies down on that side (Injury, poisoning and procedural complications) | 0 | 1
Throbbing sensation at the site of the right scalp incision (Injury, poisoning and procedural complications) | 0 | 1
Aching pain over the middle 3 fingers and palm of the right hand (Nervous system disorders) | 0 | 1
Vibration at the top left end of the ipg (Product Issues) | 0 | 1
Pollakiury (Renal and urinary disorders) | 1 | 0
Esophageal irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (upper respiratory tract infection) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The original study planned to enroll 60 subjects from a minimum of 8 sites. The study enrolled 9 patients from 3 sites. Recruitment was prematurely stopped due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No